CLINICAL TRIAL: NCT03425617
Title: Effects of Dual Bronchodilator Treatment (Tiotropium + Olodaterol Respimat) on Cardiopulmonary Interactions in Hyperinflated Patients With COPD
Brief Title: Effects of Dual Bronchodilator Treatment on Cardiopulmonary Interactions in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Dr. J. Alberto Neder, Clinical professor, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6018318
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tiotropium + Olodaterol first (Experimental): tiotropium 5 mcg plus olodaterol 5 mcg via Respimat® single dose in Visit 3 followed by PLACEBO via Respimat® single dose in Visit 4
  Interventions: Drug: Tiotropium + Olodaterol; Other: PLACEBO
- PLACEBO FIRST (Experimental): Placebo via Respimat® single dose in Visit 3 followed bytiotropium 5 mcg plus olodaterol 5 mcg via Respimat® single dose in Visit 4
  Interventions: Drug: Tiotropium + Olodaterol; Other: PLACEBO

INTERVENTIONS:
Drug: Tiotropium + Olodaterol — tiotropium 5 mcg plus olodaterol 5 mcg via Respimat® single dose
  Other Names: INSPIOLTO®
Other: PLACEBO — PLACEBO via Respimat® single dose

SUMMARY:
The deleterious consequences of lung hyperinflation seem not to be restricted to the respiratory system in patients with chronic obstructive pulmonary disease (COPD). Cardiac function, in particular, is strongly influenced by changes in lung volumes and intra-thoracic pressures. In this context, strategies to reduce lung hyperinflation and the work of breathing can positively impact upon cardiac output and blood flow redistribution to peripheral muscles in these patients. There is growing evidence that combination of bronchodilators of different classes is an efficacious and safe strategy for further improving airflow obstruction and hyperinflation in patients with more advanced COPD. Therefore, we aim to investigate that, compared with placebo, a novel LABA/LAMA fixed combination (tiotropium 5 mcg plus olodaterol 5 mcg via Respimat® (Inspiolto®) (TIO/OLO) would decrease lung volumes at rest and during exercise, thereby improving: 1) central and peripheral hemodynamics and 2) arterial oxygenation, with positive consequences on skeletal muscle oxygenation and exercise tolerance in hyperinflated patients with moderate to very severe COPD.

DETAILED DESCRIPTION:
Prospective, proof-of-concept, single-dose study will be conducted using a randomized, double-blind, placebo-controlled, crossover design. Treatment will consist of a single dose of tiotropium 5mcg and olodaterol 5mcg via Respimat (Inspiolto)(TIO/OLO) or placebo; the order of treatment will be randomized. Submaximal cardiopulmonary exercise tests will be performed 1 hour after inhalation of TIO/OLO or placebo. Changes in blood flow index (BFI) measured by near-infrared spectroscopy (NIRS) during exercise will be the primary study endpoint.

Written informed consent will be obtained from all participants prior to performing any study related procedures. Participants will complete: 1) an initial visit to determine eligibility for the study; 2) a run-in visit conducted after 2 weeks of stabilization on short-acting bronchodilator therapy to familiarize subjects with the standardized exercise test (submaximal cardiopulmonary exercise tests) to be used in the subsequent treatment visits; and 3) two treatment visits, randomized to order, conducted 3-7 days apart.

Visit 1 will include:

1. A thorough medical history;
2. Clinical assessment;
3. Chronic activity-related dyspnea evaluation;
4. Complete pulmonary function testing;
5. A symptom-limited incremental exercise test on a cycle ergometer to determine maximal exercise capacity (Wmax); and
6. Post-salbutamol pulmonary function testing for assessment of bronchodilator responsiveness.

Visit 2 will consist of discontinuous submaximal cardiopulmonary exercise testing for familiarization.

Visits 3 and 4 will consist of pulmonary function tests (spirometry, plethysmography), followed by administration of TIO/OLO or placebo. One hour after inhalation, subjects will perform pulmonary function tests (spirometry, plethysmography) followed immediately by the submaximal cardiopulmonary exercise tests.

Procedures Pulmonary function testing: Routine spirometry, body plethysmography, single-breath diffusing capacity of the lung for carbon monoxide (DLCO), and maximum inspiratory/expiratory mouth pressures will be performed according to recommended techniques using automatic equipment (Vmax 229d with Vs62j body plethysmograph; SensorMedics, Yorba Linda, CA). Measurements will be expressed as % of predicted normal values.

Cardiopulmonary exercise testing: Exercise tests will be conducted on an electronically-braked cycle ergometer using a cardiopulmonary exercise testing system (Vmax229d; SensorMedics) in accordance with clinical exercise testing guidelines. Incremental exercise testing at Visit 1 will consist of a steady-state resting period, followed by followed by 1 minute of loadless pedalling, then 10 watt increases in work-rate every minute to the point of symptom-limitation. Maximal work rate (Wmax) will be defined as the highest work rate that the subject is able to maintain for at least 30 seconds. Constant work rate testing will be conducted at all subsequent visits (see below). Measurements will be collected at rest and during exercise while subjects breathe through a mouthpiece and a low-resistance flow transducer with nasal passages occluded by a noseclip. Measurements will include: standard cardiorespiratory, metabolic and breathing pattern parameters collected on a breath-by-breath basis and compared with predicted normal values based on age and height; heart rate by 12-lead electrocardiogram; blood pressure by auscultation; dynamic operating lung volumes derived from IC maneuvers; oxygen saturation (SpO2) by pulse oximetry; arterialized blood gases from earlobe samples; the intensity of perceived leg discomfort and exertional dyspnea rated by the modified 10-point Borg scale. Breath-by-breath measurements will be averaged every 20-seconds throughout exercise. Three main time points will also be evaluated: rest will be defined as the steady-state period after at least 3 minutes of breathing on the mouthpiece while seated at rest on the cycle ergometer before exercise starts (cardiopulmonary parameters will be averaged over the last 20-sec of this period and resting ICs will be collected while breathing on the same circuit immediately after completion of the quiet breathing period); isotime will be defined as the longest duration achieved during all constant load exercise tests, and; end-exercise will be defined as the last 30-sec of loaded pedaling at the 75%Wmax stage (i.e., Tlim).

Submaximal cardiopulmonary exercise tests: constant work rate testing will consist of a steady-state resting period, followed by two stages at unloaded exercise for 5 min and 75% of Wmax to the limit of tolerance (Tlim. min).

Cardiac output and muscle blood flow and deoxygenation: Cardiac output will be assessed continuously by a calibrated signal-morphology impedance cardiography system (PhysioFlow; Manatec Biomedical, France). Near-infrared spectroscopy (NIRS; OxyMon MK III, Artinis Medical Systems, The Netherlands) will be used to evaluate skeletal muscle blood flow and deoxygenation. The optode will be placed laterally over the mid-third of the right vastus lateralis. Deoxy-hemoglobin (HHb) has been selected as a proxy for muscle fractional O2 extraction and expressed relative to maximum values elicited by cuff-induced ischemia. The NIRS system measures indocyanine green (ICG) concentration following a bolus injection of 5 mg of ICG into a forearm vein. ICG injections will be performed during the fourth minute of each exercise stage (unloaded and 75%of maximal work load).

Symptom evaluation. Dyspnea (respiratory discomfort) will be defined as the "sensation of breathing discomfort" and leg discomfort as "the sensation of leg discomfort experienced during pedalling." These sensations will be rated at rest, every minute during exercise and at end-exercise using the modified 10-point Borg scale. Upon exercise cessation, subjects will be asked to verbalize their main reason for stopping exercise, i.e., breathing discomfort, leg discomfort, combination of breathing and leg discomfort or some other reason to be specified.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years;
2. Male or female gender;
3. Long-term history of active smoking;
4. Signs and symptoms of COPD with adequate treatment according to the GOLD recommendations for at least 3 months (1);
5. A modified MRC dyspnea score ≥2 or a Baseline Dyspnea Index ≤8;
6. Resting lung hyperinflation as demonstrated by inspiratory capacity <80% predicted or functional residual capacity >120% predicted at Visit 1;
7. Objective evidence of dynamic hyperinflation (a decrease in inspiratory capacity from rest >200 mL)(24,25) and peak exercise dyspnea (breathing discomfort) ≥ leg discomfort scores during the incremental cardiopulmonary exercise test at Visit 1;
8. A positive "volume" response (≥200 mL increase in inspiratory capacity) to a bronchodilator (400μg salbutamol) at Visit 1
9. Ability to perform all study procedures and provide/sign informed consent.

Exclusion Criteria:

1. Asthma or other concomitant pulmonary disease;
2. Use of oral steroids in the preceding month;
3. Orthopedic/rheumatological limitation precluded cycling;
4. Type I or non-controlled type II diabetes mellitus or other endocrine diseases;
5. Unstable angina, life-threatening cardiac arrhythmias, use of an implantable defibrillator;
6. Myocardial infarction within the previous 6 months;
7. History of long QT syndrome (or prolonged corrected QT interval (>450 ms during screening);
8. Clinically significant ECG abnormality;
9. History of exercise-induced syncope;
10. Any contraindication for exercise testing;
11. Inability to understand and cooperate with the procedures.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Blood Flow Index (BFI) | 1 day
  Near infrared spectroscopy (NIRS)-derived muscle ICG difference divided by the rise time from 10 to 90% of peak.

SECONDARY OUTCOMES:
Cardiac output | 1 day
  Cardiac output measured by thoracic cardioimpedance
Muscle oxygenation | 1 day
  Deoxy-hemoglobin (HHb) has been selected as a proxy for muscle fractional O2 extraction and expressed relative to maximum values elicited by cuff-induced ischemia.
Tlim | 1 day
  Exercise tolerance during hugh intensity constant load exercise test (75% of peak workload)
Exercise dyspnea | 1 day
  Borg score rated during isotime and peak exercise
Inspiratory capacity | 1 day
  Inspiratory capacity, inspiratory reserve volume measured at rest, isotime and peak exercise
Inspiratory reserve volume | 1 day
  Inspiratory reserve volume measured at rest, isotime and peak exercise

CONTACTS AND LOCATIONS:
Overall Officials: J Alberto Neder, Prof, Principal Investigator — Queen'sUniversity/Kingston General Hospital
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided